CLINICAL TRIAL: NCT04146129
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 1 Single Ascending Dose Study to Assess the Safety, Pharmacokinetics, and Pharmacodynamics of CDX-0159 in Healthy Subjects
Brief Title: A Phase 1 Study of CDX-0159
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celldex Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDX0159-01
Record Dates: First submitted 2019-10-29; First posted 2019-10-31 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Healthy Subjects
Keywords: CDX-0159
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CDX-0159 (Experimental): Eligible subjects will receive a single dose of CDX-0159
  Interventions: Drug: CDX-0159
- Normal saline (Placebo Comparator): Subjects assigned to receive placebo will receive a single dose of normal saline
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: CDX-0159 — Single dose of one of four dosages of CDX-0159
  Arms: CDX-0159
Drug: Normal saline — Single infusion of normal saline
  Arms: Normal saline

SUMMARY:
This is a study to determine the safety of CDX-0159 in healthy subjects.

DETAILED DESCRIPTION:
CDX-0159 is a humanized monoclonal antibody that binds to a protein called KIT that is expressed on mast cells.

This study will evaluate the safety, pharmacokinetics, and pharmacodynamics of CDX-0159 in healthy subjects.

ELIGIBILITY:
Key Inclusion Criteria:

* An informed consent signed and dated by the subject.
* Healthy volunteer aged 18-55.
* In generally good health and without significant medical conditions based on physical exam, ECG, and laboratory test results.
* Body mass index (BMI) ≥ 18.5 kg/m2 to ≤ 30 kg/m2
* No medication other than mild analgesics, vitamins and mineral supplements or, oral contraceptives
* Both males and females of child bearing potential must agree to use a medically accepted contraceptive regimen during study and up to 150 days afterwards.
* Not a current smoker (or regular user of any nicotine containing product).
* Willing to follow all study rules

Key Exclusion Criteria:

* Women who are pregnant or nursing
* History of anaphylaxis, food allergies, or allergies (chronic or seasonal) requiring prescription medication
* Autoimmune disorders requiring more than topical medication
* History of asthma requiring the use of inhaled medication within the past 5 years.
* Vaccination with live vaccines within 4 weeks prior to study drug administration (subjects must agree to avoid vaccination during the study).
* Positive urine test for alcohol and drugs of abuse.

Other Protocol defined inclusion and exclusion criteria could apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-10-29 (Actual); Primary Completion 2020-04-06 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by CTCAE v5.0 | Day 1 to Day 43.
  Safety of single, ascending doses of CDX-0159 as determined by percentage of participants with adverse events as assessed by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Altasciences Clinical Kansas, Inc., Overland Park, Kansas, United States